CLINICAL TRIAL: NCT04165434
Title: Effect of Eight-week Concurrent Training on Functional Capacity, Force, Balance in Patients With Unilateral Transtibial Amputation
Brief Title: Effect of Eight-week Concurrent Training on Functional Capacity in Patients With Unilateral Transtibial Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Amputados
Record Dates: First submitted 2019-10-11; First posted 2019-11-18 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2018-02

CONDITIONS: Amputation of Lower Limb Above Knee; Sequelae
Keywords: Concurrent Training; Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Untrained unilateral transtibial amputees who underwent the assessment and recommended training.
  Interventions: Other: Concurrent Training
- Control (No Intervention): Untrained unilateral transtibial amputees who after the evaluation were not included for the recommended training.

INTERVENTIONS:
Other: Concurrent Training — Strength training and interval aerobic training in the same training session
  Arms: Experimental

SUMMARY:
OBJECTIVES: To assess the effect of concurrent training (CT) of an eight-week on strength, power and cardiorespiratory fitness on muscle condition, balance, load distribution in the lower limbs and aerobic capacity in patients with unilateral transtibial amputation (UTA). MATERIAL AND METHODS: Twenty-six individuals with prosthesis over 3-months were selected. Patients were randomly divided into two groups. Group 1 (n = 17) denominated UTA who performed the evaluation and training recommended by the prosthesis (bodybuilding vs. aerobic interval-training on the exercise cycle ergometer). Group 2 (n = 9) denominated untrained unilateral transtibial (UUT) amputees who after the evaluation were not included for the recommended training. All patients were evaluated at the baseline time of randomization and eight weeks after

DETAILED DESCRIPTION:
OBJECTIVES: To assess the effect of concurrent training (CT) of an eight-week on strength, power and cardiorespiratory fitness on muscle condition, balance, load distribution in the lower limbs and aerobic capacity in patients with unilateral transtibial amputation (UTA). MATERIAL AND METHODS: Twenty-six individuals with prosthesis over 3-months were selected. Patients were randomly divided into two groups. Group 1 (n = 17) denominated UTA who performed the evaluation and training recommended by the prosthesis (bodybuilding vs. aerobic interval-training on the exercise cycle ergometer). Group 2 (n = 9) denominated untrained unilateral transtibial (UUT) amputees who after the evaluation were not included for the recommended training. All patients were evaluated at the baseline time of randomization and eight weeks after. The evaluation consisted of anamnesis (inclusion criteria), clinical and functional evaluation, cardiopulmonary exercise testing, isokinetic knee testing, static and dynamic posturography. The age of the group was 28.5 ± 7.1 years old, BMI 25 ± 4.8 kg.m-2, amputation time 22 ± 27.5 months, 83% were men and 57% with amputation on the left side, 11% used antidepressants and 11% antihypertensive medicine.

KEYWORDS: Transtibial amputation; Concurrent training; Rehabilitation, Comparative Study.

ELIGIBILITY:
Inclusion criteria

* Transtibial amputation (any etiology)
* Age between 18 - 50 years
* Absence of any musculoskeletal and/or inflammatory diseases; central and/or peripheral neuropathy; psychiatry alteration
* Discharge of the rehabilitation program and the use of a prosthesis for three or more months and more.

Exclusion criteria

* Pain or inability to complete any of the tests
* High blood pressure (over 130 x 90 mmHg) before strength evaluation
* Loss of three consecutive training sessions and no return for the reevaluation session

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Functional assessment- Sit to Stand | This measure will be performing before and after the innervation (8 weeks of concurrent training 3 times a week.).
  Dynamic functional capacity assessment: patient sit to stand from a standard chair (40 centimeters high, 45 centimeters wide and backrest 90 degrees). Have to do the task five times as fast as possible time; measured in time - seconds (sec).
Functional Mobility - Time-up and Go Test | This measure will be performing before and after the innervation (8 weeks of concurrent training 3 times a week.).
  Time-up and Go Test (TUGT) - patient sit in a standard chair (40 centimeters high, 45 centimeters wide and backrest 90 degrees), trunk resting on backrest, after a verbal command has to stand up, walk for three meters (m) turn, return and sit in the chair as fast as possible; measured in time - seconds (sec).
Abiliity Test- Climb Steps | This measure will be performing before and after the innervation (8 weeks of concurrent training 3 times a week.).
  Time to climb 15 steps (height 15 centimeters / depth 30 centimeters), as quickly as possible; measured in time - seconds (sec).
Muscular strength- Isokinetic Dynamometry | This measure will be performing before and after the innervation (8 weeks of concurrent training 3 times a week.).
  Evaluation of muscular strength improvement - Isokinetic dynamometry will be use to determine knee extension and flexion strength using the Biodex Multi-Joint System 3 (Biodex MedicalTM, Shirley, NY, USA). The isokinetic variables used were maximum peak torque corrected for body weight (%), and total work (J).
Exhaled gas analyze - Ergospirometry | This measure will be performing before and after the innervation (8 weeks of concurrent training 3 times a week.).
  An exercise bike exercise test (Biocycle 2600 Electromagnetic Moviment, Brazil) was performed using the modified Astrand protocol which recommends a speed of 60 revolutions per minute (rpm) with progressive load increase (w). Two minutes (min) and the load was increased by 25 by 25 watts (w) in a stepwise fashion until maximum effort was achieved. Exhaled gas analysis was performed using the computerized metabolic gas analyzer (CPX / Ultima, MedGraphics®, St. Paul, Minnesota, USA). The maximum oxygen uptake (VO2max in ml / kg / min) was mainly evaluated.
Dynamic and static balance-Balance platform | This measure will be performing before and after the innervation (8 weeks of concurrent training 3 times a week.).
  Static and dynamic balance was evaluated by the Balance Master System version 8.1 (NeuroCom International, Inc. Clackamas, OR). The system consists of a dual force platform coupled to a microcomputer. Platform force sensors measure ground reaction force (° / s) while performing tasks such as sitting and rising from a chair by measuring the force distribution between the lower limbs in percent (%). The variables will be the mean weight transfer index (%), mean movement time (s) and mean impact index.

CONTACTS AND LOCATIONS:
Locations (1):
- Julia Maria D'Andrea Greve, São Paulo, Brazil